CLINICAL TRIAL: NCT04802746
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, 3-Way Crossover (Part A) and 2-Arm Parallel Group (Part B) Study to Assess the Pulmonary Safety of Staccato Alprazolam in Healthy Study Participants (Part A) and in Study Participants With Mild Asthma (Part B)
Brief Title: A Study to Assess the Pulmonary Safety of Staccato Alprazolam in Healthy Study Participants and in Study Participants With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0099
Record Dates: First submitted 2021-03-03; First posted 2021-03-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Healthy Study Participants; Participants With Mild Asthma
Keywords: Healthy Study Participants; Staccato alprazolam; Phase 1; Pulmonary Safety; Alprazolam; STAP-001; Mild asthma
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: Part A of the Study will be 3-Way Crossover Design and Part B will be a Parallel Design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Sequence ABC in Part A (Experimental): Study participants randomized to this arm will receive Staccato Placebo (A) and two fixed doses of Staccato alprazolam Dose 1 (B) and Staccato alprazolam Dose 2 (C) at pre-specified time points during 3 separate Treatment Periods in Part A.
  Interventions: Drug: Alprazolam; Other: Placebo
- Sequence BCA in Part A (Experimental): Study participants randomized to this arm will receive Staccato alprazolam Dose 1 (B), Staccato alprazolam Dose 2 (C), and Staccato Placebo (A) at pre-specified time points during 3 separate Treatment Periods in Part A.
  Interventions: Drug: Alprazolam; Other: Placebo
- Sequence CAB in Part A (Experimental): Study participants randomized to this arm will receive Staccato alprazolam Dose 2 (C), Staccato Placebo (A), and Staccato alprazolam Dose 1 (B) at pre-specified time points during 3 separate Treatment Periods in Part A.
  Interventions: Drug: Alprazolam; Other: Placebo
- Sequence ACB in Part A (Experimental): Study participants randomized to this arm will receive Staccato Placebo (A), Staccato alprazolam Dose 2 (C), and Staccato alprazolam Dose 1 (B) at pre-specified time points during 3 separate Treatment Periods in Part A.
  Interventions: Drug: Alprazolam; Other: Placebo
- Sequence BAC in Part A (Experimental): Study participants randomized to this arm will receive Staccato alprazolam Dose 1 (B), Staccato Placebo (A), and Staccato alprazolam Dose 2 (C) at pre-specified time points during 3 separate Treatment Periods in Part A.
  Interventions: Drug: Alprazolam; Other: Placebo
- Sequence CBA in Part A (Experimental): Study participants randomized to this arm will receive Staccato alprazolam Dose 2 (C), Staccato alprazolam Dose 1 (B), and Staccato Placebo (A) at pre-specified time points during 3 separate Treatment Periods in Part A.
  Interventions: Drug: Alprazolam; Other: Placebo
- Staccato alprazolam in Part B (Experimental): Study participants randomized to this arm will receive Staccato alprazolam at pre-specified time points in Part B.
  Interventions: Drug: Alprazolam
- Staccato placebo in Part B (Placebo Comparator): Study participants randomized to this arm will receive Staccato placebo at pre-specified time points in Part B.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alprazolam — Study participants will receive Staccato alprazolam Dose 1 and Staccato alprazolam Dose 2 at pre-specified time points in Part A. Study participants will receive single dose of Staccato alprazolam at pre-specified time points in Part B.
  Other Names: UCB7538
  Arms: Sequence ABC in Part A; Sequence ACB in Part A; Sequence BAC in Part A; Sequence BCA in Part A; Sequence CAB in Part A; Sequence CBA in Part A; Staccato alprazolam in Part B
Other: Placebo — Study participants will receive Staccato placebo at pre-specified time points in Part A and Part B matching the pre-specified Staccato alprazolam dosing.
  Other Names: PBO
  Arms: Sequence ABC in Part A; Sequence ACB in Part A; Sequence BAC in Part A; Sequence BCA in Part A; Sequence CAB in Part A; Sequence CBA in Part A; Staccato placebo in Part B

SUMMARY:
The purpose of the study is to assess the pulmonary safety of Staccato alprazolam in healthy study participants and in and study participants with mild asthma

ELIGIBILITY:
Inclusion Criteria:

Part A: Healthy study participants

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent form (ICF)
* Participants are overtly healthy at Screening and on Day -1 of each Treatment Period as determined by medical evaluation including medical history and physical examination
* Participant has a body weight of at least 45 kg (female) and 50 kg (male) and body mass index (BMI) within the range 18 to 35 kg/m^2 (inclusive)
* Participants may be male or female A male participant must agree to use contraception during the Treatment Periods and for at least 7 days after the last dose of study treatment and must refrain from donating sperm during this period

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Periods and for at least 30 days after the last dose of study treatment

* Participant is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in protocol
* Participant has normal spirometry at Screening as demonstrated by forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) ≥ 90% of predicted. In case of an out-of-range result, 1 repeat test will be allowed. If the readings are out-of-range again, the study participant will be excluded

Part B: Study participants with mild asthma

* Participant must be 18 to 55 years of age inclusive, at the time of signing the ICF
* Participant has a documented history of mild asthma diagnosed at least 6 months prior to the Screening Visit in accordance with the Global Initiative for Asthma (GINA) Guidelines 2020 and/or the National Asthma Education and Prevention Program (NAEPP) Expert Panel Report 3 Guidelines 2007. The diagnosis of mild asthma can be documented by various sources of medical information including, but not limited to, the participant's medical record, prescriptions of asthma treatments, and/or previous spirometry assessments (including FEV1 reversibility after short-acting beta2-agonist (SABA) administration)
* Participant has been on a stable asthma drug regimen (as needed short-acting beta2-agonist (SABA)s or combination low dose inhaled corticosteroids (ICS)-formoterol and maintenance treatment with daily low dose ICS or daily leukotriene receptor antagonists) for at least 4 weeks before the Screening Visit
* Participant has normal breathing sounds during normal tidal breathing on lung auscultation
* Participant has a percent predicted forced expiratory volume in 1 second (ppFEV1) value at Screening ≥80%. Before performing spirometric assessments at Screening, a washout period of at least 6 hours is required after the last SABA intake and is extended to at least 18 hours after the last intake of the combination low dose ICS-formoterol. In case of an out-of-range result, 1 repeat test will be allowed. If the readings are out of range again, the study participant will be excluded

Exclusion Criteria:

Part A: Healthy study participants

* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Participant has had a positive test for Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) or clinical signs/symptoms consistent with coronavirus disease 2019 (COVID-19) such as fever, persistent cough, shortness of breath, fatigue, and loss or change to senses of smell or taste during the 4 weeks prior to Screening or Day -1 of the first Treatment Period.
* Participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) or comparative drugs (and/or an investigational device) as stated in this protocol
* Participant has a known hypersensitivity to albuterol or similar short-acting beta2-agonist (SABA) that may be used as rescue medication administered in response to potential bronchospasm
* Participant has a history of acute narrow angle glaucoma, hydrocephalus, or Myasthenia gravis
* Participant has received or intends to use any prescription or nonprescription medicines, including enzyme inhibitors or inducers, over the counter remedies, and herbal and dietary supplements (including St. John's Wort) up to 2 weeks or 5 half-lives of the respective drug (whichever is longer) before the first administration of IMP and during the clinical part of the study, unless required to treat an adverse event (AE). This does not include oral contraceptives not exceeding 30 μg ethinyl estradiol or postmenopausal hormone replacement therapy or implants, patches, or intrauterine devices (IUDs)/intrauterine hormone-releasing systems (IUSs) delivering progesterone (for female study participants)
* Participant has previously participated in this study or participant has previously been assigned to treatment in a study of the medication under investigation in this study
* Participant has participated in another study of an IMP (and/or an investigational device) within the previous 30 days before Screening (or 5 half-lives, whichever is longer) or is currently participating in another study of an IMP (and/or an investigational device)
* Participant has a SpO2 measured by pulse oximetry <95% for >30 seconds at Screening and on day -1 of each Treatment Period. In case of an out-of-range result, 1 repeat test will be allowed. If the readings are out- of- range again, the study participant will be excluded
* Participant has a history or current condition characterized by airway hyperresponsiveness (eg, asthma, chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, obstructive sleep apnea, pneumothorax, etc) at Screening and on Day -1 of each Treatment Period
* Participant has contraindications for spirometry at Screening and on Day -1 of each Treatment Period (eg, history of myocardial infarction within 1 week, systemic hypotension, severe hypertension, significant atrial/ventricular arrhythmia, uncompensated heart failure, uncontrolled pulmonary hypertension, acute cor pulmonale, clinically unstable pulmonary embolism, history of syncope related to forced expiration/cough, history of cerebral aneurism, brain surgery within 4 weeks, recent concussion with continuing symptoms, eye surgery within 1 week, sinus surgery or middle ear surgery or infection within 1 week, presence of pneumothorax, thoracic surgery within 4 weeks, abdominal surgery within 4 weeks, late-term pregnancy, active or suspected transmissible respiratory or systemic infection, including tuberculosis within 4 weeks, physical conditions predisposing to transmission of infections, such as hemoptysis, significant secretions or oral lesions or oral bleeding; acute illness 5 days before Screening, upper respiratory tract infection in the 4 weeks before Screening)

Part B: Study participants with mild asthma

* Participant is taking a prohibited medication or has taken a prohibited medication as defined in the Protocol
* Participant has a history of or current respiratory disease characterized by airway hyperresponsiveness excluding asthma (eg, COPD, pulmonary fibrosis, obstructive sleep apnea, pneumothorax, etc)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Forced Expiratory Volume in 1 second (FEV1) to 6 hours postdose on Day 1 in Part A | From Baseline (predose Day 1) to 6 hours postdose (Day 1)
  The maximum mean treatment difference between each Staccato alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second (FEV1) will be calculated for dosing day 1 over each Treatment Period from Baseline to 6 hours postdose in Part A.
Change from Baseline in Forced Expiratory Volume in 1 second (FEV1) to 6 hours postdose on Day 4 in Part A | From Baseline (predose Day 1) to 6 hours postdose (Day 4)
  The maximum mean treatment difference between each Staccato alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second (FEV1) will be calculated for dosing days 1 and 4 over each Treatment Period from Baseline to 6 hours postdose in Part A.
Percentage of study participants with respiratory treatment-emergent adverse events (TEAEs) in Part A | From Baseline (Day 1) to Safety Follow-up period (up to Day 44)
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or comparator and events related to the procedures involved except for events in users or other persons, which only include events related to investigational devices.
Change from Baseline in Forced Expiratory Volume in 1 second (FEV1) to 6 hours postdose on Day 1 in Part B | From Baseline (predose Day 1) to 6 hours postdose (Day 1)
  The maximum mean treatment difference between each Staccato alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second (FEV1) will be calculated for dosing day 1 over each Treatment Period from Baseline to 6 hours postdose in Part B.
Change from Baseline in Forced Expiratory Volume in 1 second (FEV1) to 6 hours postdose on Day 4 in Part B | From Baseline (predose Day 1) to 6 hours postdose (Day 4)
  The maximum mean treatment difference between each Staccato alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second (FEV1) will be calculated for dosing days 1 and 4 over each Treatment Period from Baseline to 6 hours postdose in Part B.
Percentage of study participants with respiratory treatment-emergent adverse events (TEAEs) in Part B | From Baseline (Day 1) to Safety Follow-up period (up to Day 14)
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or comparator and events related to the procedures involved except for events in users or other persons, which only include events related to investigational devices.

SECONDARY OUTCOMES:
Change from Baseline in Forced Vital Capacity (FVC) to 6 hours postdose on Day 1 in Part A | From Baseline (predose Day 1) to 6 hours postdose (Day 1)
  The maximum mean treatment difference between each Staccato alprazolam dose and placebo in change from Baseline in Forced Vital Capacity (FVC) will be calculated for dosing day 1 over each Treatment Period from Baseline to 6 hours postdose in Part A.
Change from Baseline in Forced Vital Capacity (FVC) to 6 hours postdose on Day 4 in Part A | From Baseline (predose Day 1) to 6 hours postdose (Day 4)
  The maximum mean treatment difference between each alprazolam dose and placebo in change from Baseline in Forced Vital Capacity (FVC) will be calculated for dosing days 1 and 4 over each Treatment Period from Baseline to 6 hours postdose in Part A.
Change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio to 6 hours postdose on Day 1 in Part A | From Baseline (predose Day 1) to 6 hours postdose (Day 1)
  The maximum mean treatment difference between each alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio will be calculated for dosing day 1 over each Treatment Period from Baseline to 6 hours postdose in Part A.
Change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio to 6 hours postdose on Day 4 in Part A | From Baseline (predose Day 1) to 6 hours postdose (Day 4)
  The maximum mean treatment difference between each alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio will be calculated for dosing days 1 and 4 over each Treatment Period from Baseline to 6 hours postdose in Part A.
Percentage of study participants with treatment-emergent adverse events (TEAEs) in Part A | From Baseline (Day 1) to Safety Follow-up Period (up to Day 44)
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or comparator and events related to the procedures involved except for events in users or other persons, which only include events related to investigational devices.
Maximum plasma concentration (Cmax) of Staccato alprazolam in Part A | Plasma samples are collected on Day 1 and Day 4 (at Predose, and at 2 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 12 hours postdose) and on Day 2 and Day 5 (at 24 hours) of each Treatment Period.
  Cmax = maximum plasma concentration
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) of Staccato alprazolam in Part A | Plasma samples are collected on Day 1 and Day 4 (at Predose, and at 2 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 12 hours postdose) and on Day 2 and Day 5 (at 24 hours) of each Treatment Period
  AUC(0-t) = Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration
Area under the plasma concentration-time curve from time 0 to infinity (AUC) of Staccato alprazolam in Part A | Plasma samples are collected on Day 1 and Day 4 (at Predose, and at 2 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 12 hours postdose) and on Day 2 and Day 5 (at 24 hours) of each Treatment Period
  AUC = Area under the plasma concentration-time curve from time 0 to infinity
Change from Baseline in Forced Vital Capacity (FVC) to 6 hours postdose on Day 1 in Part B | From Baseline (predose Day 1) to 6 hours postdose (Day 1)
  The maximum mean treatment difference between each Staccato alprazolam dose and placebo in change from Baseline in Forced Vital Capacity (FVC) will be calculated for dosing day 1 over each Treatment Period from Baseline to 6 hours postdose in Part B.
Change from Baseline in Forced Vital Capacity (FVC) to 6 hours postdose on Day 4 in Part B | From Baseline (predose Day 1) to 6 hours postdose (Day 4)
  The maximum mean treatment difference between each alprazolam dose and placebo in change from Baseline in Forced Vital Capacity (FVC) will be calculated for dosing days 1 and 4 over each Treatment Period from Baseline to 6 hours postdose in Part B.
Change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio to 6 hours postdose on Day 1 in Part B | From Baseline (predose Day 1) to 6 hours postdose (Day 1)
  The maximum mean treatment difference between each alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio will be calculated for dosing day 1 over each Treatment Period from Baseline to 6 hours postdose in Part B.
Change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio to 6 hours postdose on Day 4 in Part B | From Baseline (predose Day 1) to 6 hours postdose (Day 4)
  The maximum mean treatment difference between each alprazolam dose and placebo in change from Baseline in Forced Expiratory Volume in 1 second/forced vital capacity (FEV1/FVC) ratio will be calculated for dosing days 1 and 4 over each Treatment Period from Baseline to 6 hours postdose in Part B.
Percentage of study participants with treatment-emergent adverse events (TEAEs) in Part B | From Baseline (Day 1) to Safety Follow-up Period (up to Day 14)
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or comparator and events related to the procedures involved except for events in users or other persons, which only include events related to investigational devices.
Maximum plasma concentration (Cmax) of Staccato alprazolam in Part B | Plasma samples are collected on Day 1 and Day 4 (at Predose, and at 2 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 12 hours postdose) and on Day 2 and Day 5 (at 24 hours) of each Treatment Period
  Cmax = maximum plasma concentration
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-t)) of Staccato alprazolam in Part B | Plasma samples are collected on Day 1 and Day 4 (at Predose, and at 2 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 12 hours postdose) and on Day 2 and Day 5 (at 24 hours) of each Treatment Period
  AUC(0-t) = Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration
Area under the plasma concentration-time curve from time 0 to infinity (AUC) of Staccato alprazolam in Part B | Plasma samples are collected on Day 1 and Day 4 (at Predose, and at 2 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 12 hours postdose) and on Day 2 and Day 5 (at 24 hours) of each Treatment Period
  AUC = Area under the plasma concentration-time curve from time 0 to infinity

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (2):
- United States (2):
  - Up0099 101, North Dartmouth, Massachusetts
  - Up0099 102, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm